CLINICAL TRIAL: NCT03714854
Title: Study of Motor Control Mechanisms in DBS-implanted Parkinson's Disease Patients
Acronym: PARKMOTEUR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties due to the loss of the engineer in charge of the TMS
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017-A03016-47
Record Dates: First submitted 2018-10-16; First posted 2018-10-22 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation; Electroencephalography; Electromyography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep brain stimulation ON (Active Comparator): Patients will undergo every experimental tasks with their DBS stimulator in ON and OFF positions. Order of ON/OFF conditions will be counterbalanced between patients.
  Interventions: Device: transcranial magnetic stimulation
- Deep brain stimulation OFF (Placebo Comparator): Patients will undergo every experimental tasks with their DBS stimulator in ON and OFF positions. Order of ON/OFF conditions will be counterbalanced between patients.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — TMS will be delivered on the sensory-motor system and the inhibitory motor control network while patients are performing behavioral and motor tasks. Brain and muscle activity will be recorded concurrently using EEG and EMG respectively.
  Other Names: electroencephalography; behavioral tasks; electromyography

SUMMARY:
Akinesia is one of the most prominent symptom in Parkinson's Disease (PD) patients. It typically consists in a inability to initiate voluntary movement, and it affects patients' quality of life. This study aims at exploring the influence of Deep Brain Stimulation (DBS) in the quality of motor control, and particularly of voluntary movement initiation, and its neural correlates. They will be evaluated using behavioral and motor tasks together with Transcranial Magnetic Stimulation (TMS) and electrophysiology (EMG and EEG).

ELIGIBILITY:
Inclusion Criteria:

* PD patients that are monitored for the tuning of their DBS stimulator by Grenoble's Hospital.
* PD patients that are hospitalized for the tuning routine 12 months after the surgical implantation.
* Good tolerance following temporary stops of the DBS stimulator
* Affiliated to a social security system
* Mental abilities sufficient for performing the behavioral tasks (MMSE score >= 24, tested less than 6 months ago)

Exclusion Criteria:

* Patients that are concerned by articles L1121-5, L1121-6, L1121-7 and L1121-8 of French Code de la Santé Publique,
* History of psychiatric or neurological illness other than PD
* Patients that are currently excluded from an other clinical trial
* Contraindications for TMS practice
* Inability to stay seated without pain for two hours
* Pregnancy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Corticospinal excitability | 60 minutes
  Corticospinal excitability is measured trough the amplitudes of TMS-evoked motor potentials recorded on the EMG at rest, and during the behavioral and motor tasks, in the two experimental conditions (DBS stimulator ON and OFF).

SECONDARY OUTCOMES:
Cortical excitability | 60 minutes
  Cortical excitability is measured trough the amplitudes of TMS-evoked potentials recorded on the EEG at rest, in the two experimental conditions (DBS stimulator ON and OFF).
Cortico-subcortical connectivity | 20 minutes
  Cortico-subcortical connectivity will be assessed on EEG signal using paired stimulation between TMS and DBS.
Correlation between behavioral and neural responses | 60 minutes
  Behavioral outcomes (such as reaction time, performance index, etc.) will be compared with neural correlates described in outcomes 1 and 2 and 3.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de GRENOBLE ALPES, Grenoble, France